CLINICAL TRIAL: NCT06710171
Title: Filling Gaps in the PrEP Cascade: User-centered Counseling About HIV Pre-exposure Prophylaxis and Linkage to Care for Gay, Bisexual and Other Men Who Have Sex with Men
Brief Title: Filling Gaps in the HIV Pre-exposure Prophylaxis Cascade Through Counseling
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-177; EFP-1129-BNG (Other Grant/Funding Number: The Ontario HIV Treatment Network)
Record Dates: First submitted 2024-09-09; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pre-Exposure Prophylaxis (PrEP); Counseling; Sexual and Gender Minorities
Keywords: gay; men who have sex with men; bisexual; HIV PrEP; Pre-exposure prophylaxis; primary care; counseling; pilot trial; HIV prevention; sexual health
MeSH Terms: conditions — Coitus; Homosexuality; Bisexuality | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized pilot trial: healthcare providers will be randomized to either of the two arms and their clients; will then answer questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online training about counseling GBM about HIV prevention with a focus on PrEP (Active Comparator): The intervention at the user level will consist of brief counseling by the participating provider about PrEP and tailored linkage to available information resources or services. This will be delivered through healthcare providers in the intervention arm, who would have completed a 60-minute online training designed by the research team.
  The intervention consists of using a theory-informed approach to user-centered brief counselling about PrEP uptake, designed specifically to help busy front-line providers in public health, sexual health and primary care settings advance clients along the PrEP cascade (specifically, supporting clients who meet evidence-based criteria for PrEP in accepting provider recommendations to use it) and provide linkage to care for related conditions.
  Interventions: Behavioral: Counseling; Other: List of resources
- Care as usual (Other): Care as usual plus a list of available community resources related to HIV prevention and/or sexual health relevant to GBM
  Interventions: Other: List of resources

INTERVENTIONS:
Behavioral: Counseling — The intervention consists of using a theory-informed approach to user-centered brief counselling about PrEP uptake, designed specifically to help busy front-line providers in public health, sexual health and primary care settings advance clients along the PrEP cascade (specifically, supporting clients who meet evidence-based criteria for PrEP in accepting provider recommendations to use it) and provide linkage to care for related conditions.
  The intervention will be delivered to GBM through participating healthcare providers who would have completed an online training designed by the research team.
  Arms: Online training about counseling GBM about HIV prevention with a focus on PrEP
Other: List of resources — This list includes webpages which contain generic information about GBMs sexual health, PrEP, mental health, information about province-wide info lines for the general public about sexual health and/or educational resources for providers.

SUMMARY:
This study s objective is to test the acceptability and feasibility of a guide to facilitate counseling about HIV prevention, focusing on HIV pre-exposure prophylaxis (PrEP). PrEP is a medication taken by HIV-negative persons to avoid an HIV infection.

Healthcare providers (including but not limited to physicians and nurses) who see gay, bisexual and other men who have sex with men (GBM) will be randomly assigned to completing a short online training versus continuing their usual activities.

The online training consists of modules containing brief information about PrEP, and about how to address concerns and difficulties that GBM face to get PrEP and to take care of their sexual health.

The investigators will ask healthcare providers to answer questionnaires before and after the research activities take place, and a member of the research team will interview some of them at the end.

Every time a healthcare provider has a counseling session with a GBM, they will facilitate putting a research coordinator in touch with the person receiving the counseling. Those GBM will also be asked to fill out questionnaires.

These activities will take place in the province of Ontario, Canada.

DETAILED DESCRIPTION:
Our research questions are: (1) Is a training program for PrEP acceptable for healthcare providers, measured by perceived advantage of applying the recommendations learned in the program, compared to current practice? (2) Is a training program for PrEP feasible for healthcare providers, measured by intention to continue applying the recommendations after the study conclusion? And (3) What is the anticipated effectiveness of a training program at increasing the proportion of PrEP-eligible GBM and TGNC who start PrEP within one month of a counseling session with a healthcare provider, compared to passive referral to existing resources?

In this open-label cluster randomized pilot trial, the investigators will randomize consenting providers to undergo an online self-paced training on brief user-centered PrEP counseling vs only receiving a list of available resources. The goal is to enroll a range of different healthcare provider types working in both urban and suburban settings, and in different work settings. Recruitment of user-participants will be facilitated by participating providers, but done by a research coordinator.

Randomization and inclusion of provider-participants is expected to start in October 2024 and will continue through February 2025. Data collection (questionnaires and interviews) will continue beyond that period for provider-participants, as well as for user-participants whose enrolment occurs during the specified recruitment dates.

The qualitative component will explore implementation considerations from the perspective of provider-participants. The investigators will do focus groups (of approximately one hour, variable size) and offer the possibility of doing individuals interviews (of approximately 30-45 minutes) if they cannot attend the focus groups.

In the analysis stage, counts and proportions will be used to describe categorical and dichotomous variables. Mean and standard deviations or median and interquartile range will be used to describe continuous normally and non-normally distributed variables respectively. For the anticipated effectiveness outcome, the intra-cluster correlation coefficient (ICC) among patient-participants will be calculated. For that purpose, our analysis will be a generalized linear mixed model (GLMM) with logit link to estimate the effect of using the training program on the probability of user-participants starting (or re-starting) PrEP, while accounting for clustering of user-participants within the respective providers.

ELIGIBILITY:
Eligible participants at the provider level ('provider-participants') will be nurses, nurse practitioners, counselors and physicians working at sexual health clinics, public health clinics and primary care practices, with or without experience giving PrEP counseling.

1A. Inclusion criteria for provider-participants:

* For practicing health-care professionals, hold a valid license to practice in Ontario (this includes resident physicians)
* Anticipate encountering a minimum of five PrEP-eligible GBM and TGNC eligible for PrEP in the three months after enrolling in the study

  1B. Exclusion criteria for provider-participants
* Anticipate to stop working at their current practice site before the end of the study

  2A. Inclusion criteria for user-participants
* Be > 19 years of age
* Self-identify as a gender different from cisgender woman
* Be presenting to their provider for sexual health/HIV testing or any other services
* Not having used PrEP in the three months prior to enrollment
* Having clinical indication for PrEP as per the Canadian PrEP guideline (i.e.: -
* Report having condomless anal sex with a man in the preceding 6 months plus any of the following: syphilis in the past year, rectal gonorrhea, LGV or chlamydia in the past year, use of PEP at least twice, ongoing sexual relationship with a person living with HIV with detectable viral load, or HIRI-MSM score > 11 if available).

  2B. Exclusion criteria for user-participants
* User-participants who have already received an invitation to participate in the study and declined will not be included since that means they would have received the intervention or the control in the past.
* Users who request getting on PrEP due to high self-perceived risk despite not meeting the clinical criteria specified above, will not be included.
* Not being able to communicate in English

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders different from cisgender woman
Enrollment: 200 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Acceptability | At the 3-month follow up of participating healthcare providers. Contextual information will be obtained using qualitative interviews (to take place within a month after the 3-month follow up)
  Proportion of provider-participants who indicate they believe using the recommendations of the training program is no different, somewhat better or significantly better than their current practice, measured with a Likert scale.

SECONDARY OUTCOMES:
Feasibility - trialability | At the 3-month follow up of participating healthcare providers. Contextual information will be obtained from of qualitative interviews, which will take place within one month after the 3-month follow up.
  Proportion of provider-participants who indicate they are somewhat likely or very likely to use the recommendations of the training program in the future, measured with a Likert scale
Feasibility - complexity | At the 3-month follow up of participating healthcare providers. Contextual information will be obtained from of qualitative interviews, which will take place within one month after the 3-month follow up.
  Ease of use of the training package (using a Likert scale). Answering somewhat easy or very easy.
Feasibility - recruitment | Measured at baseline
  Number of providers consenting to participate during the planned enrollment period (October to January)
Feasibility - retention | At the 3-month follow up of participating healthcare providers
  Proportion of provider-participants retained in the study after three months, out of provider-participants who start the training
Anticipated effectiveness | At the patient level, after each counseling session and at the 1 month follow up
  Proportion of user-participants who start (or re-start) PrEP within one month after the initial encounter

OTHER OUTCOMES:
Cost | Immediately after the completion of the online training and at the 3-month follow up of participating healthcare providers
  Additional time per patient needed to apply the intervention (numeric, in minutes)
Appropriateness | At the 3-month follow up of participating healthcare providers
  Alignment with values and culture of providers (4-point Likert scale): answering somewhat well or very well.
Fidelity | At baseline and after one month
  Degree to which the intervention was used as intended.:
  Fidelity will be measured with (1) and (2)
  1. A checklist filled out by the provider-participant during the appointments.
  2. Equivalent questions in the post-appointment questionnaire for user-participants.
  This list consists of: asking about values, addressing information gaps, talking about mental health and talking about the GBMs ability to obtain PrEP.
  The fidelity outcome will be measured by the proportion of providers indicating that they covered at least one of the topics/users indicating the providers discussed at least one of the recommended topics.
Accepting a referral to a PrEP provider | At the patient level, after each counseling session (within 5 days) and at the 1 month follow up
  Proportion of user-participants who accept a referral for PrEP
Willingness to start PrEP | At the patient level, after each counseling session (within 5 days) and at the 1 month follow up
  Change in willingness to start (or re-start) PrEP (0-10 numeric rating scale) A positive difference of one unit or higher indicating increased willingness
Perceived impact | At the 3-month follow up of participating healthcare providers
  Perceived impact (in terms of increasing the proportion of users who start PrEP) of using the intervention (4-point Likert scale): answering somewhat positive; or significantly positive impact
Satisfaction | At the patient level, after each counseling session (within 5 days) and at the 1 month follow up
  User-participant satisfaction with the clinical encounter (5-point Likert scale) Measured by the proportion of GBM indicating they were satisfied or very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Darrell H.S. Tan, MD, FRCPC, PHD, Principal Investigator — St. Michael's Hospital
Locations (1):
- Options Lab, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will be stored at St. Michael's hospital, a research and teaching site which hosts trainees at different levels working in various research projects. Data collected in this study will be used to support various research activities (abstracts, publications, presentations) by the research team and future trainees.

REFERENCES:
- See also: Current projects at Options Lab — https://optionslab.ca/projects/